CLINICAL TRIAL: NCT05007795
Title: Test to Treat TB: Impact of Sputum Sequencing-guided Individualised Therapy on Outcomes in Drug-resistant Tuberculosis (TB): a Proof of Concept Randomized Controlled Trial
Brief Title: Test to Treat TB: Impact of Sputum Sequencing-guided Individualised Therapy on Outcomes in Drug-resistant Tuberculosis
Acronym: T3-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: University of Stellenbosch (Other); Ospedale San Raffaele (Other); Stichting Katholieke Universiteit (Other); University of Cape Town Lung Institute (Other)
Responsible Party: Principal Investigator, Keertan Dheda, Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: T3-RCT; 743-2018 (Other: University of Cape Town Human Research Ethics Committee)
Record Dates: First submitted 2021-08-13; First posted 2021-08-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Tuberculosis, Multidrug-Resistant
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Programmatic MDR TB treatment regimen (No Intervention): Conventional MDR-TB laboratory tests. Sputum culture (and smear microscopy) will be evaluated monthly during the treatment period (and 6 monthly during the follow-up period) for the conventional arm.
- Sequence based resistance testing and individualized treatment (Experimental): Sputum extracted for targeted sequencing and drug resistance profile provided to clinician for individualized treatment.
  Interventions: Diagnostic Test: Targeted sequencing using the GenoScreen Deeplex assay

INTERVENTIONS:
Diagnostic Test: Targeted sequencing using the GenoScreen Deeplex assay — Targeted sequencing to be performed on DNA extracted directly from clinical sputum samples using an on-demand strategy to generate a drug resistant profile. Clinicians treating the patients will have access to this and prescribe 5 or more effective drugs to the patients within 14 days of diagnosis.
  Arms: Sequence based resistance testing and individualized treatment

SUMMARY:
Resistance to anti-tuberculosis drugs is a continually growing problem. Multidrug-resistant tuberculosis (MDRTB) is resistance to at least rifampicin and isoniazid, and extensively drug-resistant TB is additional resistance to a fluoroquinolone and a second injectable line drug. Methods currently employed in testing for resistance are inadequate and a contributing factor to the 40-50% MDR-TB treatment success rate. Current drug susceptibility testing methods are slow for most drugs, taking weeks. Rapid molecular methods such as the line probe assays, e.g. Hain GenoType MDRTBplus and sl, provide resistant calls to only a limited number of drugs, and are often less useful in smear negative patients.

Molecular technologies such as sequencing can provide a comprehensive readout of drug resistance and are able to detect resistant populations at very low levels (≤1%), thus enabling individualized therapy. This can be done directly from sputum. Targeted sequencing amplifies regions of genomic DNA associated with resistance prior to sequencing. Rapid analytic software is used to process the raw sequence data, identify resistance causing mutations and provide a readout of clinically relevant information. However, the feasibility, and more importantly the impact, of this approach has not been evaluated in a clinical trial to establish proof of concept.

Aim 1: To conduct a randomised controlled trial to determine the impact of sputum-based targeted sequencing in detecting resistance to second-line TB drugs compared to the current programmatic standard of care (Hain MDRTBplus/sl and adjunct phenotypic drug susceptibility testing) when used to inform of treatment for MDR-TB.

Aim 2: To compare currently available drug resistant sequencing pipelines for diagnostic accuracy, sensitivity, specificity and predictive value as compared to culture based phenotypic drug susceptibility testing.

Aim 3: To compare the feasibility, accuracy, turn-aroundtime, and cost implications of the above-mentioned diagnostic approaches.

DETAILED DESCRIPTION:
Trial aims:

Aim 1: To conduct a randomised controlled trial to determine the impact of sputum-based targeted sequencing in detecting resistance to second-line TB drugs compared to the current programmatic standard of care (Hain MDRTBplus/sl and adjunct phenotypic drug susceptibility testing) when used to inform of treatment for MDR-TB.

Sub-aim 1.1: To determine the proportion of patients (in the control and conventional groups) placed on ≥ 5 likely effective drugs within 14 days of rifampicin resistant tuberculosis diagnosis (the current WHO guideline) in the two groups (targeted sequencing versus LPA and phenotypic testing).

Sub-aim 1.2: To determine time-specific treatment-related outcomes (6, 12, and 18-20 month favourable outcome rates), amplification of drug resistance rates (number of drugs), and 6-month change in chest radiograph disease scores in the two groups.

Sub-aim 1.3: To determine the prevalence of minority hetero-resistant bacterial populations in patients in the same two groups and the change in these populations during the course of treatment.

Aim 2: To compare currently available drug resistant sequencing pipelines for diagnostic accuracy, sensitivity, specificity and predictive value as compared to culture based phenotypic drug susceptibility testing.

Aim 3: To compare the feasibility, accuracy, turn-around-time, and cost implications of the above-mentioned diagnostic approaches.

Patient population:

Stage 1 of this multistage study will recruit 100 patients (Stage 2 and 3 will only be undertaken if the primary outcome has been achieved in the stage 1 study). Patients aged > 18 years with newly diagnosed pulmonary rifampicin resistant tuberculosis will be recruited from the two study recruiting sites. Both HIV-infected and un-infected patients will be eligible for participation.

Study staff will be referred newly diagnosed, rifampicin-resistant cases by the staff from City of Cape Town TB Clinics and TB-specific hospitals (after a discussion with the patients) at each site. Once the patient's diagnosis has been disclosed by the attending TB doctor, the study team will meet the patient after they have commenced treatment. The study staff will screen the potential participants for eligibility to participate in the study according to the following criteria:

Inclusion criteria:

Subjects are required to meet ALL of the following inclusion criteria to participate:

* Newly diagnosed culture and/or Xpert/MTB Ultra positive pulmonary TB
* Rifampicin resistance detected using GeneXpert
* Provide written informed consent prior to all trial-related procedures
* Male or female aged 18 years and older.
* Patients on TB treatment for less than or equal to 7 days.
* Patients receiving both the shorter and longer MDR-TB regimen will be eligible.

Exclusion criteria:

Subjects will be excluded from participation if they meet ANY of the following criteria:

* A subject who in the opinion of the investigator is unlikely to cope with regular visits to the trial site either because of travel constraints, or drug or alcohol abuse, or other reason.
* Currently on MDR-TB treatment and completed 7 days of treatment.
* Any participant with a clinically significant pre-existing medical condition that, in the opinion of the investigator, may be significantly worsened by the patient's participation in the study
* Any subject with a Karnofsky score < 50.
* Having participated in other clinical studies within 8 weeks prior to trial start where investigational agents were used that may potentially impact current trial outcome.
* Participant who is pregnant, breast-feeding (and not willing to stop), or planning to conceive a child within 6 months of cessation of treatment.
* Any pre-existing laboratory abnormality, which in the opinion of the investigator will place the participant at risk (see detailed protocol for grade of abnormality).

All inclusion and no exclusion criteria must be met prior to enrolment and randomisation. Whenever the investigator has reason to suspect that there might be a health problem (other than TB), participation should only be considered after discussing the case with the medical monitor.

Trial design:

An open-label pragmatic proof of concept randomized controlled trial will be undertaken.

This will be a multi-arm multi-staged (MAMS) trial with three stages. We have funding to currently complete stage 1, but further funding will be made available through the MRC AMR EMU (PI= K Dheda) if the primary outcomes are achieved.

Stage 1 primary outcome measure: Proportion of patients initiated on treatment with ≥5 likely effective drugs within 14 days of rifampicin resistant tuberculosis diagnosis in each group (n=100).

Stage 2 primary outcome measure: Six-month unfavourable outcome rates in each group (n=230 inclusive of stage 1 patients).

Stage 3 primary outcome measure: End of treatment (12 or 18-20 month depending on the regimen used) unfavourable outcome rate in each group (n=280 inclusive of stage 2 patients)

Enrolled participants will be randomised 1:1 (open-label) to receive either the empiric standard of care (9-11 month or sometimes the 18-20 month conventional treatment regimen) or the individualised interventional regimen for MDR-TB.

Treatment duration in the conventional arm will be 9-11 months, or 18-20 months, based on the SA Department of Health Policy Guidelines for the treatment of MDR, with sputum culture (and smear microscopy) being evaluated monthly during the treatment period (and 6 monthly during the follow-up period). In the interventional arm sputum culture (and smear microscopy) will also be evaluated monthly during the treatment period (and 6 monthly during the follow-up phase).

Interventional arm:

The regimen in the interventional arm will be individualised and constructed in accordance to the Xpert/MTB Ultra, and results from targeted genome sequencing. The regimen will be developed using drugs from the table below (new WHO classification). The duration of treatment will be in accordance to the National TB program (NTP) guidelines i.e. patients who have been exposed to second-line drugs for >1 month previously, patients who require substitution of a key drug (i.e bedaquiline, linezolid or levofloxacin), those with a haemoglobin of < 8g/dl, or patients with complicated extra-pulmonary TB (meningitis, bone and complicated abdominal TB), will receive the longer regimen (18-20 months with some medications like bedaquiline and linezolid being prescribed for ~ 6 months) while all other patients will receive the NTP recommended shorter regimen (9-11 months with some medications, like bedaquiline (6 months) and linezolid (2 months), being used for shorter duration).

Note: The SA guidelines for the management of MDR-TB are currently finalised but may change slightly or over time; our study will adopt the final decision from the NTP with regards to selection/indications for the long vs. short course regimen and their respective duration of treatment.

WHO Grouping Group A: Include all three medications (unless they can not be used) - Bedaquiline, Linezolid, Levofloxacin Group B: Add both medicines (unless they cannot be used) - Clofazimine, Cycloserine/ Terizidone Group C: Add to complete the regimen and when medicines from Group A and B cannot be used - PZA, Delaminid, Ethambutol, Imipenem-cilastin/ Meropenem, Amikacin/ Streptomycin, High dose Isoniazid, Ethionamide/ Prothionamide, p-aminosalicylic, Terizidone

Conventional Arm:

Treatment in the conventional arm will be in accordance to the National TB program's recommendations. Patients on short and long course regimen will be included.

Conventional regimen for adult MDR-TB as per the SA Department of Health Policy Guidelines on the treatment of MDR:

DRUGS:

Bedaquiline (Bdq) 6 months Daily dosing Linezolid (Lzd) Only 2-months Daily Levofloxacin Daily Clofazimine Daily PZA Daily Ethambutol Daily High dose INH Daily

The conventional arm is adopted from the NTP. Any changes by the NTP to the standard of care will be mirrored in the conventional arm.

Study endpoints:

* Primary Endpoint: feasibility and impact of targeted genome sequencing to initiate more than or equal to five effective TB drugs within 14 days of diagnosis (reference standard phenotypic DST). Feasibility is a co-primary endpoint.
* Secondary efficacy endpoints:

  * favourable outcome rate (time-specific 6, 12, 18, 24 month post treatment initiation)
  * time-specific rate of treatment failure
  * time-specific culture conversion rates
  * time-specific relapse rate (including the 6 and 12 months of follow-up)
  * time-specific rates of resistance amplification
  * adverse event rates
  * cost effectiveness

Sample size calculations:

We estimate that the proportion of patients receiving effective treatment (at least 5 drugs started within 14 days) will be ~47% and ~82% in the conventional and intervention arms, respectively (rounded off conservatively to 50% and 80%; see Table 4 below for a summary readout representing detailed drug-specific calculations based on published data from several seminal studies(1-5)). Individualized therapy in the intervention arm, based on appropriate sequencing readouts, and the availability of susceptibility readouts for ethambutol and pyrazinamide will greatly reduce ineffective drugs and allow effective alternatives to be used.

Based on the assumptions outlined in Table 5, a sample size of 100 patients will allow us to detect a 30% difference in the primary outcome between the arms assuming 95% confidence, and 80% power, considering a 10% loss to follow-up rate, and an additional 1% allowance for interim analysis (performed after 50 patients are recruited). We feel that a 30% difference is what would be required to be meaningful clinically in terms of outcome relative to resource investment. We have designed a multistage trial and the sample size calculations for the stages to determine the six-month favourable outcome rate, and six-month culture conversion rate, and twelve-month favourable outcome rate are shown in Table 5.

Trial duration:

Both arms will recruit 1:1 with the duration of treatment being 9-11 months (or 18-20 months), regardless of the arm that the participant may be assigned to. The follow up will be a total duration of 12 months for both arms after treatment completion.

Ethical and management considerations:

(i) Informed consent will be obtained from all patients. The consent form will be translated into the relevant local languages and interpreters made available where necessary. Data will be kept confidential and password-protected, with all personal identifiers removed from research-related information. The patients will be given the option to withdraw from the study at any time. Pregnant patients will not be enrolled. There will be no gender bias during the conduct of the study. This study will not discriminate against HIV-infected persons and will recruit both HIV-infected and uninfected persons. Newly diagnosed HIV-infected participants will be commenced on ARV treatment using either nevirapine or a lopinavir/ritonavir combination with two other NRTI's (for compatibility with bedaquiline). HIV-infected participants already on alternative ARV treatment regimens will be changed to the above-mentioned regimen.

(v) Participants whose MDR-TB treatment has failed: In the conventional arm, management of failed MDR-TB treatment will be as per the NTP guidelines (with guidance from the provincial and national committees). In the interventional arm, participants where treatment has failed will be referred to the NTP and presented at the provincial and national committees with recommendations based on the extended DST pattern.

(vi) Management of cases of relapse and re-infection in either treatment arm: As per cases with treatment failure.

Insurance for research-related injuries:

Provided by the University of Cape Town's No-Fault Insurance

ELIGIBILITY:
Inclusion Criteria:

Subjects are required to meet ALL of the following inclusion criteria to participate:

* Newly diagnosed culture and/or Xpert/MTB Ultra positive pulmonary TB
* Rifampicin resistance detected using GeneXpert
* Provide written informed consent prior to all trial-related procedures
* Male or female aged 18 years and older.
* Patients on TB treatment for less than or equal to 7 days.
* Patients receiving both the shorter and longer MDR-TB regimen will be eligible.

Exclusion Criteria:

Subjects will be excluded from participation if they meet ANY of the following criteria:

* A subject who in the opinion of the investigator is unlikely to cope with regular visits to the trial site either because of travel constraints, or drug or alcohol abuse, or other reason.
* Currently on MDR-TB treatment and completed 7 days of treatment.
* Any participant with a clinically significant pre-existing medical condition that, in the opinion of the investigator, may be significantly worsened by the patient's participation in the study
* Any subject with a Karnofsky score < 50.
* Having participated in other clinical studies within 8 weeks prior to trial start where investigational agents were used that may potentially impact current trial outcome.
* Participant who is pregnant, breast-feeding (and not willing to stop), or planning to conceive a child within 6 months of cessation of treatment.
* Any pre-existing laboratory abnormality, which in the opinion of the investigator will place the participant at risk (see detailed protocol for grade of abnormality).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Impact of targeted genome sequencing to initiate more than or equal to five effective TB drugs within 14 days of diagnosis (reference standard phenotypic DST). | 14 days
  Impact of sputum-based targeted sequencing in detecting resistance to second-line TB drugs using the GenoScreen Deeplex assay compared to the current programmatic standard of care (Hain MDRTBplus/sl and adjunct phenotypic drug susceptibility testing) when used to inform of treatment for MDR-TB.

SECONDARY OUTCOMES:
Feasibility of targeted sequencing to initiate more than or equal to five effective TB drugs within 14 days of diagnosis. | 14 days
  To determine the proportion of patients in the interventional group with a drug-resistant profile and placed on ≥ 5 likely effective drugs within 14 days of rifampicin resistant tuberculosis diagnosis.

OTHER OUTCOMES:
Favourable outcome rate | 6, 12, 18, 24 month post treatment initiation
  Rate of favourable outcome (cure or treatment complete) in conventional and interventional arms
Rate of treatment failure | 6, 12, 18, 24 month post treatment initiation
  Rate of treatment failures in conventional and interventional arm
Culture conversion rates | 6, 12, 18, 24 month post treatment initiation
  Culture conversion rates in conventional and interventional arm
Relapse rate | 6 and 12 months of follow-up
  Rate of relapse in conventional and interventional arm
Rates of resistance amplification | 12 and 24 months post treatment initiation
  Rates of resistance amplification in conventional and interventional arm
Adverse event rates | 6, 12, 18, 24 month post treatment initiation
  Adverse event rates in conventional and interventional arm
Cost effectiveness | 24 month post treatment initiation
  Cost implications of the targeted sequencing diagnostic approach compared to the current programmatic standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Keertan Dheda, MD/PhD, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available to researchers who provide methodologically sound proposals to the principal investigator.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months to 5 years following publication.
Access Criteria: Individual participant data will be made available to researchers who provide methodologically sound proposals beginning 3 months and ending 5 years following publication. Data sharing requests should be directed to keertan.dheda@uct.ac.za. A data access agreement will need to be concluded.